CLINICAL TRIAL: NCT03844672
Title: Impact of E-cigarette Characteristics on Reinforcement and Tobacco Use Patterns Among
Brief Title: Impact of E-cigarette Characteristics on Reinforcement and Tobacco Use Patterns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tracy Smith, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 00081069; K01DA047433 (NIH)
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Smoking; Tobacco Use
MeSH Terms: conditions — Smoking; Tobacco Use | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Concentration / Low Power (Experimental): Participant will receive an e-liquid with a low nicotine concentration and an e-cigarette with a low power for three weeks.
  Interventions: Behavioral: Low Power; Behavioral: Low Concentration
- Low Concentration / High Power (Experimental): Participant will receive an e-liquid with a low nicotine concentration and an e-cigarette with a high power for three weeks.
  Interventions: Behavioral: High Power; Behavioral: Low Concentration
- High Concentration / Low Power (Experimental): Participant will receive an e-liquid with a high nicotine concentration and an e-cigarette with a low power for three weeks.
  Interventions: Behavioral: Low Power; Behavioral: High Concentration
- High Concentration / High Power (Experimental): Participant will receive an e-liquid with a high nicotine concentration and an e-cigarette with a high power for three weeks.
  Interventions: Behavioral: High Power; Behavioral: High Concentration

INTERVENTIONS:
Behavioral: Low Power — Participants will receive a low power e-cigarette to use for 3 weeks
  Arms: High Concentration / Low Power; Low Concentration / Low Power
Behavioral: High Power — Participants will receive a high power e-cigarette to use for 3 weeks
  Arms: High Concentration / High Power; Low Concentration / High Power
Behavioral: Low Concentration — Participants will receive a low concentration e-liquid to use for 3 weeks
  Arms: Low Concentration / High Power; Low Concentration / Low Power
Behavioral: High Concentration — Participants will receive a high concentration e-liquid to use for 3 weeks
  Arms: High Concentration / High Power; High Concentration / Low Power

SUMMARY:
The purpose of this project is to understand how different e-cigarettes influence their likeability and use among current smokers who try using e-cigarettes. Participants will receive an e-cigarette to sample over a three week period. During this time period they will complete daily electronic diaries and weekly lab visits. The results from this information will help understand how different types of e-cigarettes are likely to influence cigarette and e-cigarette use.

ELIGIBILITY:
Inclusion criteria include

* adults who have been smoking daily
* interested in using e-cigarettes
* who have a smartphone that can receive text messages and access to the internet or has an e-mail account that they check daily

Exclusion criteria include

* minimal prior e-cigarette use
* use of tobacco products other than cigarettes
* current use of cessation medications
* pregnant, trying to become pregnant, or breastfeeding,
* recent history of cardiovascular distress in the last three months (e.g., arrhythmia, heart attack, stroke, uncontrolled hypertension),
* household member currently enrolled in the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Smith, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Concentration / Low Power | Low Concentration / High Power | High Concentration / Low Power | High Concentration / High Power
Started | 23 | 24 | 23 | 23
Completed | 17 | 18 | 17 | 15
Not Completed | 6 | 6 | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Concentration / Low Power | Low Concentration / High Power | High Concentration / Low Power | High Concentration / High Power | Total
Number analyzed (Participants) | 23 | 24 | 23 | 23 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (12.0) | 48.9 (13.3) | 51.3 (13.1) | 49.7 (11.2) | 49.7 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 12 | 12 | 48
  Male | 10 | 13 | 11 | 11 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 4 | 4 | 13
  White | 19 | 22 | 19 | 17 | 77
  More than one race | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Cigarettes Per Day
Description: Participants complete weekly surveys reporting the number of cigarettes smoked each day on a continuous scale
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Low Concentration / Low Power | Low Concentration / High Power | High Concentration / Low Power | High Concentration / High Power
Number analyzed (Participants) | 18 | 21 | 17 | 17
cigarettes per day | 13.1 (9.3) | 12.6 (6.0) | 12.2 (8.8) | 13.3 (9.3)

2. Secondary Outcome: Average Number of E-cigarette Puffing Episodes
Description: Participants complete weekly surveys reporting the number of e-cigarette puffing episodes each day on a continuous scale
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Low Concentration / Low Power | Low Concentration / High Power | High Concentration / Low Power | High Concentration / High Power
Number analyzed (Participants) | 18 | 21 | 17 | 17
cigarettes per day | 4.8 (5.4) | 6.5 (10.7) | 5.4 (4.5) | 3.0 (4.0)

3. Secondary Outcome: Number of Choices to Smoke Cigarette in Lab Setting
Description: Participants complete lab-based choice task at Week 3 visit in which they choose between smoking conventional cigarette and e-cigarette over 10 trials. Outcome is number of times each participant chooses to smoke conventional cigarette.
Time Frame: Week 3
Measure: Mean (Standard Error); unit: Events
Arm/Group | Low Concentration / Low Power | Low Concentration / High Power | High Concentration / Low Power | High Concentration / High Power
Number analyzed (Participants) | 18 | 21 | 17 | 17
Events | 1.7 (0.42) | 2.4 (0.38) | 1.8 (0.44) | 2.4 (0.43)

ADVERSE EVENTS:
Time Frame: Two months
Arm/Group | Low Concentration / Low Power | Low Concentration / High Power | High Concentration / Low Power | High Concentration / High Power
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 12/23 | 13/24 | 12/23 | 11/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Concentration / Low Power (N=23) | Low Concentration / High Power (N=24) | High Concentration / Low Power (N=23) | High Concentration / High Power (N=23)
Headache (Nervous system disorders) | 2 (2) | 5 (5) | 4 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (6) | 3 (3) | 1 (1)
Increased Phlegm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (3)
Throat and Mouth Irritation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Burning in the Throat (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (2)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Lung Problems (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT03844672/Prot_SAP_000.pdf